CLINICAL TRIAL: NCT03939871
Title: Phase II Study of Fluvestrant Combined With Oral Vinorelbine in Hormone Receptor-positive Advanced Breast Cancer
Brief Title: A Study of Fluvestrant Combined With Oral Vinorelbine in Hormone Receptor-positive Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1564
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Hormone Receptor Positive Advanced Breast Cancer
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Fluvestrant in combination with oral Vinorelbine Fluvestrant: administered at a dose of 0.5g once im every 28 days. Vinorelbine: administered at a dose of 60mg/kg once a week for 3 weeks p.o. every 28 days.
  Interventions: Drug: fluvestrant + oral vinorelbine

INTERVENTIONS:
Drug: fluvestrant + oral vinorelbine — Eligible patients will be treated with the fluvestrant + oral vinorelbine regimen until the disease progresses or intolerable toxicity
  Other Names: there is no other intervention name

SUMMARY:
This is a single-center phase II study designed to evaluated the efficacy and safety of fulvestrant in combination with oral vinorelbine in hormone receptor-positive advanced breast cancer

DETAILED DESCRIPTION:
This is a single-group, single-center phase II trial. Patients with hormone-receptor-positive, Her2-negative recurrent or metastatic breast cancer who had not previously received any systemic antitumor therapy for advanced disease were treated with fulvestrant combined with oral vinorelbine as a first-line regimen. Key issues to be addressed in this study: to observe and evaluate the efficacy and safety of fulvestrant combined with oral vinorelbine in the treatment of hormone-receptor-positive and HER2-negative advanced breast cancer. Thirty patients are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 year-old women; Pathologically or cytologically confirmed breast cancer; Hormone receptor-positive
* ECOG score: 0-1, expected survival time ≥ 3months;
* Recurrence after adjuvant therapy or metastatic breast cancer and chemotherapy naïve in the metastatic setting or had one prior regimen for metastatic breast cancer.
* Patients must have measurable disease according to RECIST criteria Version 1.1. Bone metastases lesions were excluded.
* The patients have adequate hematologic and organ function.

Exclusion Criteria:

* Patients with symptomatic brain metastases.
* Patients who are known or suspected to be allergic to the active ingredient or excipients of the investigational drug.
* Received ≥1 standard chemotherapy regimen (excluding endocrine therapy) for advanced breast cancer.
* Participation in other clinical trials within 4 weeks before enrollment.
* Severe cardiovascular disease, including history of congestive heart failure, acute myocardial infarction within 6 months before enrollment, transmural myocardial infarction measured by ECG, uncontrolled arrhythmia, angina requiring therapy, clinically significant valvular heart disease, uncontrolled hypertension.
* Severe or uncontrolled infection.
* Any factors that affect the oral administration and absorption of drugs (such as inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.);
* Active malignancy in the past 5 years (other than carcinoma in situ of the cervix or basal cell carcinoma of the skin).
* Patients who are pregnant , breastfeeding ,or refuse to use adequate contraception during the course of participation.
* Need to concurrent other cancer therapy(other than palliative care for non-target lesions).
* Other ineligible conditions according to the researcher's judgment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-12 (Actual); Primary Completion 2020-12-12 (Estimated); Study Completion 2020-12-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | approximately 1.5 years
  PFS will be defined as the time from first dose of study drug until documentation of disease progression or death from any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | approximately 6 months
  The ORR will be calculated as the proportion of patients in the Efficacy Evaluable patient Set who achieve complete response (CR) and partial response (PR)
Incidence and Severity of adverse events | approximately 1.5 years
  hematologic toxicity，hepatotoxicity and so on

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cacner Center/ Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China